CLINICAL TRIAL: NCT03607500
Title: Effect of Moderate Caloric Restriction on Glomerular Growth After Kidney Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Abhijit Naik, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00134686; P30DK089503 (NIH)
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Kidney Transplant; Complications; Glomerular Disease; Weight Gain; Kidney Transplant
Keywords: Caloric Intake Reduction; Dietician
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caloric Intake Reduction (Experimental): The intervention group will be seen by the kidney disease dietician at all clinical visits for the first 3 months (weekly for month 1, every other week for months 2 and 3). During months 2 and 3, in the weeks that the patients are not in clinic, they will receive telephone calls from the dietician. Thus the intervention involves weekly assessment for the first 3 months (in person or over the telephone). After 3 months, the patient will not receive any further active dietary intervention from the dieticians unless the patient wishes to continue using the dieticians advice per clinic protocol.
  Interventions: Behavioral: caloric intake reduction
- Standard of care (No Intervention): The standard of care arm will receive dietary guidance per current University of Michigan Transplant Center policy, where a one time face-to-face visit is provided in the first month after kidney transplant and then as requested by the patient or referred by physician.

INTERVENTIONS:
Behavioral: caloric intake reduction — The caloric intake reduction arm will been seen by the kidney disease dietitian at all clinical visits for the first 3 months (weekly for month 1, every other week for months 2 and 3).
  Arms: Caloric Intake Reduction

SUMMARY:
One possible reason that weight gain after transplant may interfere with new kidney function is due to the enlargement of a kidney structure called the glomerulus.

The researchers believe that modest caloric intake reduction (CIR) early after kidney transplantation can reduce the enlargement (hypertrophy) of the glomerulus associated with kidney transplantation and may improve long term allograft survival, by reducing glomerular hypertrophy mediated progressive glomerulosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of kidney transplants where a post perfusion biopsy is obtained
* Body Mass Index between 25-30 kg/m2 at the time of randomization
* Non-diabetic
* Have a smart phone or active internet connection at home

Exclusion Criteria:

* Patients on dual anti platelet agents or are on oral anti coagulation medication
* Patients who have had Bariatric Surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Naik, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caloric Intake Reduction | Standard of Care
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one participant was involved in the entire trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Caloric Intake Reduction | Standard of Care | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Change in Baseline and 3 Month Glomerular Volume Between the Intervention and the Control Arm
Time Frame: Post-Perfusion (Time 0 or Study Enrollment) and 3 months
Population: Because only one participant was involved in the entire trial, showing data could violate privacy interests. Further since the outcome measure was to compare the intervention against a control, given that there is no control arm, such a comparison is impossible.
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Difference in the Number of Glomerular Ki67 Positive Cells Between the Intervention and the Control Arm
Description: 3 month protocol biopsies will be stained with monoclonal antibodies against Ki67 to identify actively dividing cells and counted manually.
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Difference in the Number of Glomerular DAPI Positive (Nuclei) Between the Intervention and the Control Arm
Description: 3 month protocol biopsies will be stained with monoclonal antibodies against DAPI to identify nucleated cells in the glomerulus and counted manually.
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Difference in the Number of TLE4 Positive (Podocyte Nuclei) Between the Intervention and the Control Arm
Description: 3 month protocol biopsies will be stained with monoclonal antibodies against TLE4 to identify podocytes and counted manually.
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Differences in Podocyte Detachment Rate Between the Intervention and the Control Arm
Description: Urine samples obtained at the time of 3-month protocol biopsies will be utilized to compare the urinary podocin mRNA to urinary creatinine ratio
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Difference in the Podocyte Hypertrophic Stress Between the Intervention and the Control Arm
Description: Urine samples obtained at the time of 3-month protocol biopsies will be utilized to compare the urinary podocin mRNA to nephrin mRNA ratio
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Difference in Glomerular Filtration Rate (GFR) at 3 and 12 Months Between the Intervention and the Control Arm
Description: Differences in glomerular filtration rate (GFR) using both creatinine (modified diet in renal disease) as well as serum cystatin C based equations
Time Frame: 3 months, 12 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Difference in Proteinuria Between the Intervention and the Control Arm
Description: Proteinuria measured by laboratory samples
Time Frame: Measured through study completion, about 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Difference in Glycosylated Hemoglobin (HbA1c) Percent in the Intervention and the Control Arms
Description: Measure the difference in HbA1c between the two arms during 3 month protocol biopsies
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Difference in Weight of Participants in the Intervention and Control Arms
Description: Weight as measured by pounds
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Caloric Intake Reduction | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through each participant's study completion, typically 3 months
Description: Participant had no SAEs or AEs and outlived the trial.
Arm/Group | Caloric Intake Reduction | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT03607500/Prot_SAP_000.pdf